CLINICAL TRIAL: NCT04347603
Title: Sedation or General Anesthesia During Trancatheter Aortic Valve Implantation Procedure : ANESTAVI Study
Brief Title: Sedation or General Anesthesia During TAVR
Acronym: ANESTAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL19_0350; UF7825 (Other: CHU Montpellier); 2020-A00497-32 (Other: ID-RCB)
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-05

CONDITIONS: Stenoses, Aortic
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- General Anesthesia (Experimental): - General anesthesia : After pre-anesthetic preparation (25-50 mg Hydroxizine orally), the anesthesia induction will be performed by IV perfusion of Propofol 1 to 2 mg/kg, Sufentanyl for analgesia 0,2 to 0,4 µg/kg, curarisation with Atracurium 0,15 mg/kg. The anaethesia depth will be monitored by the bispectral index (BIS). Orotracheal intubation will be performed, the patient will be ventilated to controlled volume with 6-8 mL/kg of current volume based on expected body weight (PBW). The respiratory rate will be adjusted to have an ETCO2 between 35 and 45 mmHg. The anesthesia will be maintained through the Sevorane at 0.7-1 MAC, the average blood pressure will be controlled through a pressure cuff with a target between 60 and 80 mmHg. The Fio2 will be adapted to obtain saturation > 94% with 5 cmH2O PEEP.
  Interventions: Procedure: TAVR
- Local Anesthesia (Active Comparator): Local anesthesia at the device introduction site will be obtained by infiltration of Naropein.
  Interventions: Procedure: TAVR

INTERVENTIONS:
Procedure: TAVR — Femoral percutaneous aortic prosthesis (TAVR)

SUMMARY:
Transcatheter aortic valve replacement TAVR is become the reference method for patients with severe aortic stenosis who are contraindicated or at risk for surgical aortic replacement. Initially performed under general anesthesia (GA), recent developpement of minimalist approach of TAVR include the use of local anesthesia (LA) with or without conscious sedation (CS) associated with full percutaneous access and no routine transoesophageal echocardiography (T0E). The aim is to simplify the procedure and to allow fast recovery of patients with early discharge and reduced cost.

Evidence guiding the decision of whether to perform TAVR under GA or LA-CS is limited to non-randomized trials and registry data Current evidence is however limited by probable patient selection bias, methodological variability between studies, various methods of anesthesia and a lack of agreement regarding appropriate clinical end-points. The potential benefits of TAVR with LA include reduced procedure time, shorter intensive care unit (ICU) length of stay, reduced need for intraprocedural vasopressor support, and the potential to perform the procedure without the direct presence of an anesthetist for cost-saving reasons. As LA with CS is preferred with good results in main centers, GA may be useful to facilitate intraprocedural TOE which is necessary in case of intraprocedural complications and may facilitate the procedure for the physician particularly when the patient is anxious or disturbed. A resulted better concentration without precipitation may influence the outcomes in term of valve positioning. The patient comfort could also be better during femoral puncture or rapid pacing. The aim of the study is to compare transfemoral TAVR under general anesthesia (experimental group) versus local anaesthesia with sedation (control group) with a safety primary combined end point of adverse events at 72 h follow-up (hemodynamic parameters and VARC 3 criteria). Secondary end points include hospitalization length, satisfaction of the patients and operators and 30 days mortality.

The hypothesis is a non inferoirity of the GA staregy regarding the primary end point.

DETAILED DESCRIPTION:
Implantation of a femoral percutaneous aortic prosthesis (TAVI) has become a routine therapy for elderly patients with severe aortic stenosis (SA) and a high or intermediate surgical risk. With growing experience of intereventional temas with the technique, improvement of device technology, and expansion of the technique to patients with lower surgical risk, the procedure is mostly currently performed under local anaesthesia with or without conscious sedation (TAVR-LA-CS) rather than by the traditional general anaesthesia approach (TAVR-GA).

The purpose of this study is to compare the safety (primary outcome) and efficiency (secondary outcome) of local anesthesia (LA) with conscious sedation (CS) versus general anesthesia (GA) for the TAVR procedure performed with transfemoral access.

This is a blindly randomized, non-inferiority controlled trial. The study will include all consecutive patients referred to the Cardiology Department of the CHU of Montpellier, France, for TAVR by transfemoral access which is the default strategy. Procedure is indicated for severe symptomatic aortic valve stenosis with high or intermediate surgical risk or with contraindication to surgery and after decision of the multidisciplinary team according to the current recommendations of the European society of cardiology. Patients are randomized into two groups with surgical risk stratification : one with general anesthesia (experimental group) and one with local anesthesia with sedation: (control group) in a 1/1 ratio. Exclusion criteria include contraindication to GA or LA-CS based on hemodynamic status or comorbidities. The primary composite endpoint combines the major peri and post-operative adverse events (72 hours), including hemodynamic instability and major complications (VARC 3 criteria). Secondary criteria include length of intensive care unit (ICU) hospitalization and total hospital stay, duration of intervention, analgesic dose up to 72 hours, finger oximetry results, transition to GA in the AL group, fluoroscopic time, patient and operator satisfaction (questionnaires for patients, interventional cardiologists and anesthesiologists) and mortality at 30 day follow-up.

It is expected that 20% of patients will have an event defined by the main judgement outcome. To balance the various expected benefits of LA-CS over the length of stay, duration in ICUC and opioid drug use, the non-inferiority threshold was set at an absolute difference of up to 15%, or 35% of event rates in the experimental arm.

Based on this threshold and the above assumptions, and using 80% power and 5% Type I error (for a one-sided test), 109 patients are must be included in each arm, for a total of 218 patients with a randomization rate of 1:1.

The inclusion period will be 24 months or as soon as the required number of subjects is reached. Follow-up includes a medical assessment during the peri-operative period (72h) and at the end of the hospital stay and a clinical evaluation by phone survey at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Consecutive patients referred to the cardiology department of the CHU in Montpellier, France, for TAVI via transfemoral access.
* Patients for whom the procedure is indicated after decision by the heart team and according to the current recommendations of the European Society of Cardiology.
* Patients with severe aortic stenosis defined by mean gradient > 40 mmHg and/or aortic valve area 1 cm2 or 0.8 cm2/m2 as recommended. May also include patients with low gradient (< 40mm hg) and low flow (stroke volume index < 35ml/minute) which are classic indications for aortic valve replacement
* Ability to consent to participate in study
* Patient affiliated with or beneficiary of a social security scheme

Exclusion Criteria:

* Chronic respiratory insufficiency treated by long term oxygeno therapy
* Pulmonary hypertension above 50mmHg
* BMI>35
* TAVI by carotidian or apical way
* Pregnant women
* Vulnerable person according to L1121-6 of Public Health reglementation in France

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Hemodynamic instability | within 72 hours after intervention
  Hemodynamic instability (defined by the need for fluid loading >1500 ml associated or not with the use of inotrope support) within the first 72 hours
Major complications (according to VARC 3 criteria) | within 72 hours after intervention
  Major complications (according to VARC 3 criteria) within the first 72 hours :
  * death in hospital,
  * major vascular events,
  * neurological events,
  * myocardial infarction,
  * aortic regurgitation >2,
  * conductive disorders requiring pacemaker implantation,
  * acute renal failure (KDIGO criteria),
  * pericardial tamponade.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University hospital, Montpellier
  - University hospital, Nîmes

IPD SHARING:
Plan to Share IPD: Undecided